CLINICAL TRIAL: NCT06086431
Title: Dexamethasone Vs. Dexmedetomidine for Erector Spine Plane Block in Pain Management After Pediatric Idiopathic Scoliosis Surgery.
Brief Title: Dexamethasone Vs. Dexmedetomidine for ESPB in Pain Management After Pediatric Idiopathic Scoliosis Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14/2023
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-01

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis | interventions — Sodium Chloride; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): 0.2% ropivacaine for erector spinae plane block
  Interventions: Drug: 0.9% sodium chloride
- Dexamethasone (Active Comparator): 0.2% ropivacaine + 0.1mg/kg Dexamethasone for erector spinae plane block
  Interventions: Drug: Dexamethasone
- Dexmedetomidine (Active Comparator): 0.2% ropivacaine + 0.1ug/kg Dexmedetomidine for erector spinal plane block
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: 0.9% sodium chloride — administration of 0.5ml/kg of 0,2% ropivacaine + 0.01ml/kg 0.9% sodium chloride for the erector spine plane block
  Other Names: placebo
  Arms: Placebo
Drug: Dexamethasone — administration of 0.5ml/kg of 0.2% ropivacaine with 0.1mg/kg Dexamethasone for the erector spine plane block
  Arms: Dexamethasone
Drug: Dexmedetomidine — administration of 0.5ml/kg of 0.2% ropivacaine with 0.1ug/kg Dexmedetomidine for the erector spine plane block
  Arms: Dexmedetomidine

SUMMARY:
Effect of perineurial dexamethasone and dexmedetomidine on erector spinal plane block duration for pediatric, idiopathic scoliosis surgery.

DETAILED DESCRIPTION:
This study is proposed to explore the effect of perineurial Dexamethasone and Dexmedetomidine on erector spinal plane block duration for pediatric, idiopathic scoliosis surgery.

After scoliosis surgery, children need good analgesia. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anesthesia is essential in children due to the much lower toxicity threshold of local anesthetics. An effective adjuvant, such as Dexamethasone or Dexmedetomidine, could allow for a higher dilution of local anesthetics while maintaining and enhancing their analgesic effect.

There is considerable research where intravenous and perineural dexamethasone and Dexmedetomidine use has been compared in adults. However, there is a massive lack of research regarding children.

In this study, investigators compare perineural Dexamethasone and Dexmedetomidine. Group 2 has dexamethasone doses of 0.1mg/kg, and group 3 has 0,1ug/kg Dexmedetomidine added to the local anesthetic.

The investigator aims to find a dexamethasone or dexmedetomidine that covers the need for good pain relief and fast recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* children scheduled for idiopathic scoliosis surgery
* age >10 and <18 years

Exclusion Criteria:

* age < 10 years
* age < 18 years
* infection at the site of the regional blockade
* coagulation disorders
* immunodeficiency
* ASA= or >4
* steroid medication in regular use

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
first need of opiate | 48 hours
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid consumption | 48 hours
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 16 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 20 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
NLR | 24 and 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 24 and 48 hours after surgery]
  Platelet-to-lymphocyte ratio
MEP | durring surgery
  motor evoced potentials
Nerve damage [range 0-4] | 12 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 24 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 48 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
adverce effects | 48 hours after surgery
  nausea, vomitting, bradycardia, hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Kotwicki, Prof.dr hab., Study Director — Poznan University of Medical Sciences
Locations (1):
- Department of Spine Diseases and Pediatric Orthopedics, University of Medical Sciences, Poznań, Poland, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No